CLINICAL TRIAL: NCT07192536
Title: Accelerated Neuromodulation for Concurrent Post-Traumatic Stress Disorder (PTSD) & Chronic Pain in Veterans - Exploring Preliminary Efficacy and Feasibility
Brief Title: Accelerated Neuromodulation for Concurrent Post-Traumatic Stress Disorder (PTSD) & Chronic Pain in Veterans
Acronym: ANCHOR
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Legion Veterans Village Research Foundation (Other)
Responsible Party: Principal Investigator, Venugopal Karapereddy, Psychiatrist; Clinical Assistant Professor (University of British Columbia), Legion Veterans Village Research Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00083064
Record Dates: First submitted 2025-08-31; First posted 2025-09-25 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain; Post-traumatic Stress Disorder (PTSD)
Keywords: Transcranial Magnetic Stimulation (TMS); PTSD; chronic pain; Veterans; Theta burst stimulation; Brain stimulation; Neuromodulation; Military; Accelerated treatment protocol
MeSH Terms: conditions — Chronic Pain; Stress Disorders, Post-Traumatic | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This preliminary clinical study is an open label, non-randomized, single group, proof of concept design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Accelerated Neuromodulation Treatment (Experimental): Intermittent theta burst stimulation (iTBS), is a non-invasive treatment that uses brief magnetic pulses to stimulate specific areas of the brain. This treatment delivers pulses in very short bursts that mimic natural brain rhythms, and may be effective in treating Post-Traumatic Stress Disorder (PTSD) and chronic pain. Each treatment takes approximately 3 minutes to complete. In this open label, single arm study, participants will undergo an accelerated treatment schedule over a period of 5 days. On day 1, participants will receive 1-2 sessions, and on days 3-5 they will receive 5-6 sessions per day (with a 45 minute break between each iTBS session).
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Intermittent theta burst stimulation (iTBS) will be delivered via the Magstim Horizon 3.0 Transcranial Magnetic Stimulation device. This device has been authorized by Health Canada (License No.: 111334, Type: System, Device class: 3 Device first issue date 2024-06-04, License name: HORIZON 3.0 TMS THERAPY SYSTEM) and is indicated for use in treating mild depressive disorder. The device will be used off-label as a potential treatment for Post-Traumatic Stress Disorder (PTSD) and chronic pain in this Investigator-Initiated study. rTMS will be delivered using modified intermittent theta burst accelerated bilateral treatments (MITAB), combining low frequency 1HZ to the right dorsolateral prefrontal cortex (dlPFC) with high frequency intermittent theta burst to the left dlPFC, up to 6 times per day for 5 days.

SUMMARY:
The ANCHOR study is testing a novel, non-invasive brain stimulation program designed specifically for Veterans experiencing concurrent post-traumatic stress disorder (PTSD) and chronic pain. These conditions often occur together and can greatly impact daily life. Current treatments options for PTSD and chronic pain are limited, may come with severe side-effects, and often take weeks if not months to see results.

In this study, participants will receive an intensive one-week course of intermittent theta burst stimulation (iTBS), a Health Canada-approved technology already used for depression. In this study, it is being tested for its potential to reduce both PTSD and chronic pain symptoms.

This clinical trial will recruit 30 Veterans, all of whom will receive the active treatment (there is no placebo). Participants will receive 5-6 sessions of iTBS per day (each treatment lasts approximately 3 minutes) over a period of 5 days (one week total duration). Researchers will track changes in PTSD symptoms, chronic pain, mood, anxiety, daily functioning, and cognitive performance at 4 time points: baseline (before treatment), at the end of treatment ( end of week 1), and at 2 follow-up assessments (3 weeks and 6 weeks after the end of treatment).

The goal of this study is to determine whether this unique brain stimulation program is able to treat concurrent PTSD and chronic pain in Canadian Veterans. This study also aims to lay the groundwork for larger trials that could expand access to innovative treatments for the Veteran community.

DETAILED DESCRIPTION:
This is an open label, non-randomized, single group, proof of concept design study. Military Veterans experiencing concurrent PTSD and chronic pain will undergo an an intensive one-week rTMS theta burst protocol with multiple stimulation session per day. Follow-up assessments will take place 3-weeks and 6-weeks post final treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (>19years age) with symptoms of both post-traumatic stress disorder (PTSD) and chronic pain, confirmed by clinical interview and rating scales (CAPS-5 & CPGS) performed at screening visit

   a. Participants must score either 'Moderate' or 'Severe' on the CAPS-5 scale, and 'Grade I, II, or III' on the CPGS to qualify
2. Any sex and gender identity
3. Willing and able to attend all study visits and adhere to treatment plan, including the use of a personal computer to complete at-home questionnaires
4. Able to understand the informed consent form, study procedures and willing to participate in study
5. Able to perform the testing required by the study

Exclusion Criteria:

1. Exhibiting significant suicide risk, as defined by:

   1. a. suicidal ideation as indicated by items 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) within the past six months, at screening visit
   2. demonstrating suicidal behaviours or non-suicidal self-injury within the past six months, or;
   3. clinical assessment of significant suicidal risk or risk of self-injury during participant interview
2. Participants who are pregnant, nursing, or planning a pregnancy
3. Participants who engage in sexual intercourse which could result in pregnancy, and who do not agree to use a highly effective contraceptive method throughout their participation in the study
4. Any other clinically significant neurological, psychiatric, cardiovascular, pulmonary, gastrointestinal, hepatic, renal, vascular or any other major concurrent illness that, in the opinion of the Investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if he/she takes part in the study
5. Have participated in another clinical trial within the last 30 days or are currently enrolled in another interventional clinical trial
6. Individuals who have active or inactive implants (including device leads), including deep brain stimulators, cochlear implants, and vagus nerve stimulators, as well as metallic implants such as electrodes, stents, clips, pins, plates, screws, braces, or other metallic objects such as shrapnel or permanent jewelry.
7. The presence of ferrous metal pins or plates in or near the head (within 30 cm of the coil). Including implanted electrodes/stimulators, aneurysm clips or coils, stents, bullet fragments, or other implants.
8. Individuals who have history of epilepsy or unexplained seizure history.
9. Uncontrolled/severe symptomatic cardiovascular disease states including: recent myocardial infarction (within prior 6 months); history of stroke; and hypertension (resting blood pressure >150/100)
10. History of intracranial mass, intracranial haemorrhage/stroke, cerebral trauma/traumatic brain injury or increased intracranial pressure
11. Any defects in the neurocranium (e.g. after skull trepanation)
12. Skin diseases of the scalp

    Contraindications for NeuroCatch Platform:
13. Clinically documented hearing issues (e.g., in-ear hearing problems or punctured ear drum)
14. In-ear hearing aid or cochlear implant, hearing device
15. Lack of fluency in the English language
16. Unhealthy scalp (apparent open wounds and/or bruised or weakened skin)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Post-traumatic Stress Disorder Checklist for DSM-5 (PCL-5) score | Baseline to End of Treatment (end of week 1), Follow up Assessments (week 3, week 6 after nil-treatment)
  The PCL-5 is a 20-item self-report checklist of Post-Traumatic Stress Disorder (PTSD) symptoms based closely on the DSM-5 criteria. Respondents rate each item from 0 ("not at all") to 4 ("extremely") to indicate the degree to which they have been bothered by that particular symptom over the past month (or past week if using the PCL-5 weekly). A total symptom severity score (range: 0-80) can be obtained by summing the scores for each of the 20 items, with higher scores indicating more severe PTSD symptoms. A score greater than 33 is typically used to indicate severity sufficient for a PTSD diagnosis
Change in Chronic Pain Grade Scale (CPGS) score | Baseline to End of Treatment (end of week 1), Follow up Assessments (week 3, week 6 after nil-treatment)
  The CPGS assesses two dimensions of overall chronic pain severity: pain intensity and pain-related disability. It is suitable for use in all chronic pain conditions. Participants must score 'Grade I, II, or III' on the CPGS at screening to qualify for the study. Each questions is scored using a 11-point Likert scale. Total scores range from 0 to 30, with higher scores indicating more pain.
Change in Pain Disability Index (PDI) score | Baseline to End of Treatment (end of week 1), Follow up Assessments (week 3, week 6 after nil-treatment)
  The PDI is designed to measure the degree to which aspects of a participant's life are disrupted by chronic pain. In other words, how much pain is preventing them from doing what they would normally do or from doing it as well as they normally would. Participants will be asked to respond to each category indicating the overall impact of pain in their life, not just when pain is at its worst. The total PDI score can range from 0 to 70, a higher score indicating more disruption with functioning across a range of activities.

SECONDARY OUTCOMES:
Change in Hamilton Depression Rating Scale (HAM-D) score | Baseline to End of Treatment (end of week 1), Follow up Assessments (week 3, week 6 after nil-treatment)
  The Hamilton Depression Rating Scale (HAM-D) contains 17 questions which detect change and measure illness severity. Individual items are rated on a scale of 0-4, 0-3, and 0-2 with total HAM D score range from 0 (not ill) to 53 (severely ill).
Change in Patient Health Questionnaire (PHQ-9) score | Baseline to End of Treatment (end of week 1), Follow up Assessments (week 3, week 6 after nil-treatment)
  The PHQ-9 is a 9-item self-report questionnaire used to assess depression symptom severity. Depression symptoms are rated from 0 (not depression) to 27 (severe).
Change in Hamilton Anxiety Rating Scale (HAM-A) score | Baseline to End of Treatment (end of week 1), Follow up Assessments (week 3, week 6 after nil-treatment)
  The Hamilton Rating Scale for Anxiety (HAM-A) is used as a rating measure of anxiety severity. The scale consists of 14 items. Each item is rated on a scale of 0 to 4. The HAM-A total score is the sum of the 14 items and the score ranges from 0 (no anxiety) to 56 (severe anxiety)
Change in General Anxiety Disorder scale (GAD-7) score | Baseline to End of Treatment (end of week 1), Follow up Assessments (week 3, week 6 after nil-treatment)
  The General Anxiety Disorder scale is a 7-item questionnaire used to measure symptoms of generalized anxiety disorder. Scores range from 0-21 with higher scores indicating more generalized anxiety
Change in Inventory of Psychosocial functioning (IPF) score | Baseline to End of Treatment (end of week 1), Follow up Assessments (week 3, week 6 after nil-treatment)
  The IPF is a self-report instrument measuring PTSD-related functional impairment experienced by Veterans. Respondents rate how often they have acted a certain way over the past 30 days. The IPF was developed to have high content validity, to not confound PTSD symptoms and related impairment, and to not require respondent attributions regarding the cause of impairment. Items are rated on a 7-point scale ranging from 0 ("never") to 6 ("always"). The IPF yields a total score (0-66) and scores for seven subscales: romantic relationships, family, work, friendships and socializing, parenting, education, and self-care functioning (lower indicates better functioning/less impairment). Higher scores indicate more impairment
ReadON Cognitive Test | Baseline to End of Treatment (end of week 1), Follow up Assessments (week 3, week 6 after nil-treatment)
  Cognitive function, specifically executive functioning, processing speed, episodic memory, and working memory, will be assessed using the ReadON Cognitive Test (Orange Neurosciences, Kingston, ON, Canada). Unlike standardized paper tests with a single total score, the ReadON test uses an algorithm to provide a comprehensive profile across multiple cognitive domains.
NeuroCatch® Platform | From baseline visit to end of treatment visit (end of week 1)
  NeuroCatch® Platform (NCP; NeuroCatch Inc., Surrey, BC, Canada) will be used to complement as an objective measure of cognitive function. NCP is an easy-to-use, objective, rapid neuro-physiological brain function assessment system, licensed by Health Canada as a Class II medical device. The platform provides acquisition, display, analysis, storage, reporting, and management of EEG and event related potential (ERP) information including the N100, P300 and N400 measures of brain function
Program Feasibility will be assessed using the Effectiveness Framework | Through study completion, an average of 1 year
  Efficacy/effectiveness will be assessed using results from the clinician- and participant-reported Post-Traumatic Stress Disorder (PTSD) and chronic pain symptoms measured as primary outcome measures (PCL-5 and CPGS), comparing changes from baseline to end of treatment (end of week 1).
Program Feasibility will be assessed using the Adoption Framework | Through study completion, an average of 1 year
  Adoption will be assessed as the perceived ease of protocol administration (for clinicians) and program adherence (for participants).
Program Feasibility will be assessed using the Implementation and Maintenance framework | Through study completion, an average of 1 year
  Implementation and maintenance will be assessed upon qualitative reports from the study team and participants regarding barriers and facilitators to help inform future program implementation efforts

OTHER OUTCOMES:
Program Feasibility will be assessed using the Reach framework | Through study completion, an average of 1 year
  Reach will be assessed as the proportion of participants screened who are eligible for the study, reason(s) for ineligibility, number of withdrawals/dropouts, barriers to participation reported by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Venugopal Karapereddy, FRCP(C), Principal Investigator — University of British Columbia (UBC); Brainstim Health;
Locations (1):
- Brainstim Health, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No